CLINICAL TRIAL: NCT02882945
Title: Polymorphism Analysis of HLA-DRB1*04 Alleles in Patients With Type 2 Diabetic Macroangiopathy in Northeast Chinese
Brief Title: Gene Polymorphism Associated With Macroangiopathy in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Weihua Wu, Director, First Affiliated Hospital of Harbin Medical University
Other Study IDs: HarbinMU_WHW_001
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Angiopathies
MeSH Terms: conditions — Diabetic Angiopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory analysis Blood samples were collected after over-night fasting, and serum was stored at -20°C.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group A: 150 healthy blood donors without a family history of diabetes mellitus
  Interventions: Other: Group A
- Group B: 200 cases of type 2 DM without complications (group B), there were 62 males and 108 females, aged 29-53, with an average age of 42 ± 9 years
  Interventions: Other: Group B
- Group C: 120 cases of type 2 DM with macroangiopathy complication (group C), there were 70 males and 50 females, aged 40-53, with an average age of 47 ± 6 years. Among the group C subjects, 65 individuals had CHD; 55 patients had cerebrovascular disease (CVD); and 30 subjects had a combination of peripheral vascular diseases (PVD) and CHD
  Interventions: Other: Group C

INTERVENTIONS:
Other: Group A — 150 healthy blood donors without a family history of diabetes mellitus were enrolled in the study.
  Other Names: healthy blood donors
  Groups: Group A
Other: Group B — 200 cases of type 2 DM without complications were enrolled in the study.
  Other Names: type 2 DM without complications
  Groups: Group B
Other: Group C — 120 cases of type 2 DM with macroangiopathy complication were enrolled in the study.. Among the group C subjects, 65 individuals had CHD; 55 patients had cerebrovascular disease (CVD); and 30 subjects had a combination of peripheral vascular diseases (PVD) and CHD.
  Other Names: type 2 DM with macroangiopathy complication
  Groups: Group C

SUMMARY:
To explore the possible implications of HLA-DRB1*04 alleles in patients with type 2 DM and macroangiopathy

DETAILED DESCRIPTION:
Previous studies examining the molecular etiology of diabetes mellitus in China and abroad have mainly focused on the relationship between HLA and type 1 diabetes mellitus (DM) (1-3). Due to the complexity of type 2 DM heredity, few researchers have studied the correlation between type 2 DM and HLA. In recent years, it has been suggested that the development of coronary heart disease (CHD) in diabetic individuals is not merely a complication of diabetic macroangiopathy. CHD and diabetic macroangiopathy share some genetic associations. Previous studies have demonstrated that certain HLA*DRB1*04 subtypes are associated with an increased risk of cardiovascular disease.

Experimental methods: For genomic DNA extraction, 3-5ml venous blood samples were collected from all patients. Coagulation was prevented using EDTA.

The procedure for PCR amplification was as follows: denaturing for 100s at 96°C, annealing for 60s at 63°C, 1 cycle; denaturing for 10s at 96°C, annealing for 60s at 63°C, 9 cycles; denaturing for 10 s at 96°C, annealing for 30 s at 59°C; extending for 30 s at 72°C, 20 cycles; maintaining at 4°C. Analyzing PCR products stained by Ethidium Bromide on 2.5% agarose gel electrophoresis. Bands were observed using an ultraviolet light and a biological imaging system.

Statistical method: The degree of agreement with Hardy-Weinberg equilibrium was determined using the χ2 test. A t-test was employed for comparison of CRP levels (M ± s) and a χ2 test was performed to compare allelic frequencies. The relative risk rate (RR) was calculated as (Number of patients with the gene×Number of people in control group without the gene) divided by (Number of people in control group with the gene×Number of the patients without the gene). PC was calculated using Fisher's method if χ2 > 3.84.

ELIGIBILITY:
Inclusion Criteria:

* clinical CHD (such as angina pectoris, myocardial infarction) diagnosed by dynamic electrocardiogram and ultrasonic cardiogram;
* coronary atherosclerosis confirmed by coronary angiographic examination;
* cerebral infarction diagnosed by cerebral CT;
* common carotid artery intimal-media thickness (IMT) ≥1.2 mm measured by Doppler ultrasonic examination;
* extensive irregular stenosis of a lower extremity artery (diameter < 3mm) or segmentally obstructed.

Exclusion Criteria:

* age < 20 years
* age > 60 years

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 150 healthy blood donors without a family history of diabetes mellitus at the Harbin Blood Disease Research Center were enrolled in the study, and 320 outpatients and hospitalized patients of type 2 diabetes mellitus from the First and Second Affiliated Hospital of Harbin Medical University.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Test of allelic frequencies | At recruitment
  A commercially available kit was used for extraction of genomic DNA from the whole blood samples (PEL-FREEZ Inc., USA). Thirty-two pairs of sequence-specific primers (SSP) for HLA-DRB1*04 alleles were purchased from One Lambda, Inc. (USA), and the Taq enzyme was purchased from Promega Corp. (USA). The PCR-SSP technique was employed to determine the HLA-DRB1*04 alleles for each subject. Genes were amplified using the 5700 PCR thermal cycler manufactured by Applied Biosystems Inc. (USA).

SECONDARY OUTCOMES:
Evaluation of serum CRP(C-reactive protein) levels | At recruitment
  A commercially available 96-well plate ELISA assay kit (introassay CV 1.7%~3.9%, interassay CV 2.8%~5.1%) was used to quantify hs-CRP in serum (DSL Inc., USA). All samples were evaluated in duplicate. The absorbance (OD) was determined using a BIO-RAD2550 microwell plate reader (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Nan Ma, Master, Principal Investigator — First Affiliated Hospital of Harbin Medical University

IPD SHARING:
Plan to Share IPD: Undecided